CLINICAL TRIAL: NCT00578799
Title: Effects of Probiotics in Patients With Ulcerative Colitis.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Non applicable clinical trial
Sponsor: University of California, Irvine (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCRT07053 [2007-6028]
Record Dates: First submitted 2007-12-18; First posted 2007-12-21 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kyo-Dophilus (Active Comparator): Kyo-Dophilus (5x109 bacteria/capsule, twice a day, 1 in the morning, 1 in the evening)
  Interventions: Dietary Supplement: Kyo-Dophilus
- Placebo (Placebo Comparator): placebo capsules (potato starch)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Kyo-Dophilus — 5x109 bacteria/capsule, twice a day, 1 in the morning, 1 in the evening
  Arms: Kyo-Dophilus
Dietary Supplement: placebo — placebo capsules (potato starch
  Arms: Placebo

SUMMARY:
This study is being conducted in patients who have been diagnosed with ulcerative colitis (UC), a form of inflammatory bowel disease (IBD) - a disease of the intestine.

The purpose of this study is to test the therapeutic (medical treatment) effects of daily consumption of Kyo-Dophilus (a commercially available dietary supplement often used by individuals with inflammatory bowel disease) on their UC. Kyo-Dophilus consists of three probiotic bacteria (beneficial bacteria to help maintain the balance of good bacteria in the intestine) to help treat inflammatory bowel disease caused by bad bacteria. Patients will still be maintained on their clinical standard of care for their UC as part of their participation in this study.

DETAILED DESCRIPTION:
Probiotics are defined as "live microorganisms, which, when administered in adequate amounts, confer a health benefit on the host." Most probiotics are lactic acid producing bacteria that are endogenous to the human GI (gastrointestinal) tract and are commonly utilized in the fermentation of food products, such as yogurt. Disturbances in the composition of the bacterial flora of the GI tract are associated with diarrhea and inflammatory bowel disease (IBD), and consumption of some strains of probiotic bacteria are very effective for treating diarrhea and possibly individuals with ulcerative colitis (UC). We will test the effects of 3 strains of probiotic bacteria on UC. In addition to standard medical care for UC, participants will consume a dietary supplement of 3 probiotic bacteria (Kyo-Dophilus; Lacobacillus acidophilus, Bifidobacterium bifidum, and Bifidobacterium longum) for 6 weeks. Changes in clinical symptoms and physiological markers of systemic and GI inflammation in subjects with UC will be assessed. Significant effects of the probiotics will be determined by comparing pre- and post-probiotic treatment measures for disease severity and level of inflammation and by comparing the probiotic treated group with the placebo treated control group. Any placebo effect on UC will also be assessed.

Forty subjects with ulcerative colitis will be recruited for the study and be provided a dietary supplement (5x109 bacteria/capsule, twice a day) for 6 weeks to 1/2 of the subjects and 1/2 of the UC subjects will be given a placebo control (potato starch). Standard medical care and therapies will be continued throughout the study. Initially, the physician will complete the Ulcerative Colitis Disease Activity Index (UCDAI) and the participants will complete the Shortened Inflammatory Bowel Disease Questionnaire (SIBDQ), and biopsies collected for histopathological assessment and analysis of inflammatory cytokine production (mRNA). Also, 30 ml of venous blood will be collected from each subject for analysis of serum/plasma levels of inflammatory cytokines and stress hormones. Subjects will be randomly assigned to the probiotic or placebo group (blinded to the physicians). After consuming the dietary supplement or placebo for 6 weeks, subjects will complete the SIBDQ questionnaire, the physician complete the UCDAI, be examined by sigmoidoscopy and tissue biopsies and blood samples collected. Also, during the 6 weeks of treatment, subjects will maintain a daily diary of their bowel habits. Data analysis will determine whether, relative to placebo controls, consumption of probiotics reduces the symptoms and levels of intestinal inflammation in patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* We will be studying patients with mild to moderate active ulcerative colitis (UC).
* Patients are eligible to participate if:

  * they are between 18 and 65 yr of age;
  * have an endoscopic and histologic confirmed diagnosis of UC for at least 1 yr; and
  * have at least a 2 week history of active UC that has not responded to mesalamine therapy.
* Subjects will not have consumed any fermented products, such as yogurt, for at least 6 weeks prior to being entered into the trial.

Exclusion Criteria:

* Subjects will be excluded if they have the following:

  * Crohn's disease,
  * disease less than 25 cm from the anal canal,
  * active enteric infection,
  * evidence of severe disease characterized by hemoglobin <8.0 g/dl, white blood cell count >20,000 cells/mm3, temperature >38.5◦C, albumin <25 g/dl, active disease >2 months, UCDAI < 2 or >9,
  * history of dysplasia of the colon or any cancer within 5 years,
  * clinically significant hematologic values (see above) or biochemical values (serum creatinine concentrations >1.5 times the upper limit of normal or alkaline phosphatase, aspartate aminotransferase, or alanine aminotransferase concentrations >2.5 times the upper limit of normal) are also ineligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The UCDAI (Ulcerative Colitis Disease Activity Index) scores will be used to measure disease remission | 2 years
Results of patient questionnaires. | 2 years
Histopathological scoring of disease activity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dwight M Nance, Ph.D, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Health Sciences Medical Center, Orange, California, United States